CLINICAL TRIAL: NCT07012226
Title: Effects of an Energy-restricted Diet on the Expression of the Sirtuin-1 and Leptin Receptor Genes in White Blood Cells, and Cardiometabolic Markers in Individuals With Hypertriglyceridemia: Comparison Between Low and High Weight Loss Responders
Brief Title: Comparison of Cardiometabolic Markers in Individuals With Hypertriglyceridemia With Low and High Weight Loss Responses to an Energy-restricted Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate professor, Shahid Beheshti University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 43014022
Record Dates: First submitted 2025-05-27; First posted 2025-06-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Obesity and Overweight; Hypertriglyceridaemia
MeSH Terms: conditions — Obesity; Overweight; Hypertriglyceridemia | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-calorie diet (Other): Low-calorie diet
  Interventions: Other: Low-calorie diet

INTERVENTIONS:
Other: Low-calorie diet — Low-calorie diet based on calculated calorie needs

SUMMARY:
Total RNA is extracted from isolated white blood cells, and cDNA is synthesized from these samples. Subsequently, the expression levels of the SIRT1 and leptin receptor genes are determined through quantitative PCR.

DETAILED DESCRIPTION:
Hypertriglyceridemia (HTG), defined as fasting triglycerides (TGs) ≥150 mg/dL, is a prevalent condition in the adult population, with an increasing prevalence that parallels the rise in obesity rates. There is a robust body of literature indicating a correlation between mild to moderate HTG and a number of complications, including cardiovascular disease and pancreatitis.

Lifestyle changes and weight loss could improve HTG. Dietary calorie restriction is a cornerstone in the weight loss program. However, the rate of achieving substantial weight loss through dietary interventions is often not high. Consequently, identifying factors associated with responders to both desirable and undesirable weight loss before initiating dietary interventions can help individuals struggling with weight loss. In this context, gene expression markers have been proposed as promising tools. For instance, a number of studies have identified predictors of body weight and improvement in glycemic status by comparing the transcriptomic profile of adipose tissue from obese and overweight individuals during a low-calorie diet. In other studies, peripheral blood cells have been utilized for the examination of gene expression profiles. Peripheral blood cells, including white blood cells, are readily available and, express most of the human genome. Consequently, they can reflect the gene expression of key tissues affecting energy homeostasis in response to nutritional changes or weight change. Sirtuin-1 (SIRT1) gene expression, a known regulator of glucose and lipid homeostasis, is altered by caloric restriction and weight loss. It is possible that the basal level of SIRT-1 expression may predict the metabolic response to weight loss. Conversely, leptin exerts influence over several physiological processes, including communication with the central nervous system, energy expenditure, and food intake. Obese individuals may exhibit higher levels of leptin resistance and reduced access to the central nervous system via the blood-brain barrier in comparison to lean individuals. The extent of leptin receptor expression may serve as a determining factor in these disparities. Consequently, the level of leptin receptor expression may also influence the response of individuals to a weight loss program.

The present study aims to evaluate the expression of SIRT-1 and leptin receptor genes in white blood cells and changes in cardiometabolic factors in individuals with hypertriglyceridemia associated with overweight and obesity. The variables will be compared at the beginning and end of the study between those who have lost less weight after two months and those who have lost more weight. The relationship of these variables to the percentage of weight loss will also be examined. The primary hypothesis posited that specific pre-weight loss factors could predict optimal weight loss responders. Secondary hypotheses were formulated with the objective of investigating how cardiometabolic markers would be affected by weight loss in response to a hypocaloric diet in subjects with HTG.

Methods:

The study population consists of people with mild to moderate hypertriglyceridemia who are overweight or obese and are placed on a low-calorie diet program.

Inclusion criteria:

* Mild to moderate hypertriglyceridemia (TG=150-500 mg/dL)
* Body mass index (BMI) greater than 25
* Not using fibrates

Exclusion criteria:

* Advanced chronic kidney disease patients
* Patients with liver cirrhosis
* Any change in the treatment plan during the study, including changes in the type and dose of medications taken or the start of medications that affect blood lipids.

All individuals deemed eligible will be placed on a low-calorie diet. The duration of the study is 2 months. To this end, the Mifflin formula is employed to calculate the requisite calories, with the level of physical activity factored into the calculation to determine the daily calorie requirement. Subsequently, 500 calories are deducted from this figure to derive a low-calorie diet. The determination of food groups is then based on their respective caloric content, with carbohydrates assigned a value of 50% of calories and protein assigned a value of 20% of calories. Carbohydrates should be obtained primarily from foods with a low to medium glycemic index, and simple sugars (monosaccharides, disaccharides) should be strictly limited. Patients are encouraged to choose healthy fats (monounsaturated and polyunsaturated fats). The duration of the study is 2 months.

At the end of the study, participants will be divided into tertiles based on the percentage of weight loss during the two-month period. Subsequent comparisons of study outcomes will be made between tertile 1 and tertile 3.

Venous blood samples will be collected from all patients following an overnight fast in to heparinized tubes. Following the centrifugation of the whole blood sample, the plasma is initially separated and subsequently frozen until the test is conducted. Additionally, the buffy coat, which contains leukocytes and is delineated by the interface between plasma at the superior aspect and red blood cells at the inferior aspect, is separated. Subsequent to this separation, the RNA Later solution is added to the buffy coat, which is then stored in a freezer. Total RNA will be extracted from isolated white blood cells using Trizol, and cDNA will be synthesized from these samples. Subsequently, the relative expression levels of the leptin receptor and SIRT-1 genes are determined through the use of specific primers and SYBR green master mix and Step-one plus system. The plasma sample is analyzed to measure several key parameters, including the lipid profile, insulin, leptin, adiponectin, C-reactive protein, and interleukin-6, by using commercial kits. The data will undergo analysis using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hypertriglyceridemia (TG=150-500 mg/dL)
* Body mass index (BMI) greater than 25
* Not using fibrates

Exclusion Criteria:

* Advanced chronic kidney disease patients
* Patients with liver cirrhosis
* Unwillingness to continue cooperating with the study
* Any change in the treatment plan during the study, including changes in the type and dose of medications taken or the start of medications that affect blood lipids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-01-12 (Actual); Study Completion 2026-01-27 (Actual)

PRIMARY OUTCOMES:
Gene expression of SIRT1 | up to 2 months
  Expression levels of SIRT1 gene in white blood cells
Plasma lipid profile | up to 2 months
  The plasma concentrations of triglycerides, cholesterol, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol

SECONDARY OUTCOMES:
Plasma adipokines | up to 2 months
  Plasma concentrations of adiponectin, leptin, and insulin.
Gene expression of leptin receptor | up to 2 months
  Gene expression of the leptin receptor in leukocytes
Plasma inflammatory markers | up to 2 months
  Plasma concentrations of the inflammatory markers C-reactive protein and interleukin-6

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition Clinic located in the Faculty of Nutrition Sciences, Shahid Beheshti University of Medical Sciences, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No
I do not have access to a reputable external site to share IPD information.